CLINICAL TRIAL: NCT01927978
Title: Using "PET Response Criteria in Solid Tumors (PERCIST)" in Evaluating Response to Neoadjuvant Chemoradiotherpy for Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201207067MIC
Record Dates: First submitted 2013-08-15; First posted 2013-08-23 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; 18F-FDG PET; staging; therapy planning; therapy response monitoring; prognosis
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- esophageal cancer, 18F-FDG PET

SUMMARY:
This study is aimed to evaluate the effectiveness of 18F-FDG PET in the initial staging, therapy planning, and therapeutic response monitoring for esophageal cancer patients.

Purpose:

1. The incremental staging information by using 18F-FDG PET
2. The impact of the PET results on the patients' subsequent therapy planning
3. To compare treatment response using RECIST criteria and FDG PET results.

DETAILED DESCRIPTION:
Background: Esophageal cancer is one of the leading malignancies in Taiwan. Accuracy tumor staging can direct to appropriate therapy planning and provide prognostic implications. Positron emission tomography (PET) with [18F]-fluoro-2-deoxy-D-glucose (FDG) has been shown to have better N staging and prognostic stratification abilities than conventional imaging modalities, such as endoscopic ultrasonography (EUS) and CT.

Purpose: This study is aimed to evaluate the effectiveness of 18F-FDG PET in the initial staging, therapy planning, and therapeutic response monitoring for esophageal cancer patients.

Method: Patients with pathological proven esophageal cancer, age 20-90 year-old, will be included in this study. Each patient will receive a baseline PET study. For those patients who received pre-operative CCRT, another PET will be performed 1-4 weeks after completion of CCRT.

Primary outcome: 1. The incremental staging information by using 18F-FDG PET 2. The impact of the PET results on the patients' subsequent therapy planning 3. To compare treatment response using RECIST criteria and FDG PET results.

Secondary outcome: To correlate the PET response rate and the patients' disease free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Age：20-90 years old
2. Histological proved esophageal cancer
3. ECOG performance status 0-2
4. written informed consent signed

Exclusion Criteria:

1. prior chemotherapy or treatment for other systemic anti-cancer agent(s)
2. pregnant or intend to be pregnant
3. other malignancies known
4. other concurrent cancer treatment

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histological proved esophageal cancer
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-08 (Estimated); Study Completion 2014-08 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of 18F-FDG PET in the initial staging, therapy planning, and therapeutic response monitoring for esophageal cancer patients. | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yen Ruoh Fang, M.D.,Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Enzinger PC, Mayer RJ. Esophageal cancer. N Engl J Med. 2003 Dec 4;349(23):2241-52. doi: 10.1056/NEJMra035010. No abstract available. PMID 14657432
- [Background] Ng T, Vezeridis MP. Advances in the surgical treatment of esophageal cancer. J Surg Oncol. 2010 Jun 15;101(8):725-9. doi: 10.1002/jso.21566. PMID 20512949
- [Background] Chatterton BE, Ho Shon I, Baldey A, Lenzo N, Patrikeos A, Kelley B, Wong D, Ramshaw JE, Scott AM. Positron emission tomography changes management and prognostic stratification in patients with oesophageal cancer: results of a multicentre prospective study. Eur J Nucl Med Mol Imaging. 2009 Mar;36(3):354-61. doi: 10.1007/s00259-008-0959-y. Epub 2008 Oct 18. PMID 18931839
- [Background] Yen TJ, Chung CS, Wu YW, Yen RF, Cheng MF, Lee JM, Hsu CH, Chang YL, Wang HP. Comparative study between endoscopic ultrasonography and positron emission tomography-computed tomography in staging patients with esophageal squamous cell carcinoma. Dis Esophagus. 2012 Jan;25(1):40-7. doi: 10.1111/j.1442-2050.2011.01204.x. Epub 2011 May 19. PMID 21595776
- [Background] Barber TW, Duong CP, Leong T, Bressel M, Drummond EG, Hicks RJ. 18F-FDG PET/CT has a high impact on patient management and provides powerful prognostic stratification in the primary staging of esophageal cancer: a prospective study with mature survival data. J Nucl Med. 2012 Jun;53(6):864-71. doi: 10.2967/jnumed.111.101568. Epub 2012 May 11. PMID 22582047
- [Background] Yanagawa M, Tatsumi M, Miyata H, Morii E, Tomiyama N, Watabe T, Isohashi K, Kato H, Shimosegawa E, Yamasaki M, Mori M, Doki Y, Hatazawa J. Evaluation of response to neoadjuvant chemotherapy for esophageal cancer: PET response criteria in solid tumors versus response evaluation criteria in solid tumors. J Nucl Med. 2012 Jun;53(6):872-80. doi: 10.2967/jnumed.111.098699. Epub 2012 May 11. PMID 22582049